CLINICAL TRIAL: NCT03665870
Title: Prevention Through Intervention: Telehealth Solution to Deter 911 Calls Due to Hypoglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Birmingham Fire and Rescue Service (Unknown)
Responsible Party: Principal Investigator, Mohanraj Thirumalai, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UAB-CHSP-2017-1
Record Dates: First submitted 2018-08-29; First posted 2018-09-11 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus; Hypoglycemia Unawareness; Hypoglycemia; Hypoglycemia Acute
Keywords: Telehealth; Emergency Medicine; Paramedicine; Diabetes; Hypoglycemia; Telecoaching
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia

STUDY DESIGN:
Intervention Model Description: Single arm pre-post study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Hypoglycemia Education: Participants will receive educational support to prevent repeat episodes of hypoglycemia.
  Interventions: Behavioral: Hypoglycemia Education

INTERVENTIONS:
Behavioral: Hypoglycemia Education — Two in-person visits to the home of the participant and 4 phone calls will be conducted to provided education on prevention of hypoglycemia.

SUMMARY:
This study aims to standardize and evaluate the benefits of the Prevention to Intervention program offered by the Birmingham Fire and Rescue Service. This will accomplished by standardizing the educational materials used, offering phone based follow-up and pre-post data collection.

ELIGIBILITY:
Inclusion Criteria:

1. Be a citizen of Birmingham
2. Be 18 years or older
3. Receive Dextrose-50 IV (intravenous treatment provided by EMS personnel for hypoglycemia)
4. Understand and speak English

Exclusion Criteria:

a) Enrolled currently in any diabetes related educational programs

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-05-24 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Fear of Hypoglycemia | Through study completion, an average of 8 weeks
  One of the most important impact of hypoglycemia, is non-compliance to diabetes treatment due to the fear of hypoglycemia. This would be measured using the "Hypoglycemia Scale: FH-15" scale.

SECONDARY OUTCOMES:
Self Efficacy | Pre and Post (after 8 weeks)Through study completion, an average of 8 weeks
  Measured using the "Perceived Diabetes Self-Management Scale".
Knowledge of Diabetes | Through study completion, an average of 8 weeks
  Measured using the "The Knowledge in Low Literacy in Diabetes Knowledge Assessment Scale"

CONTACTS AND LOCATIONS:
Overall Officials: Mohanraj Thirumalai, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Birmingham Fire and Rescue Service, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thirumalai M, Zengul AG, Evans E. Challenges and Lessons Learned From a Telehealth Community Paramedicine Program for the Prevention of Hypoglycemia: Pre-Post Pilot Feasibility Study. JMIR Diabetes. 2021 Aug 3;6(3):e26941. doi: 10.2196/26941. PMID 34342593